CLINICAL TRIAL: NCT05976880
Title: Grip Effects of Power Ball in Children With Visual Impairment
Brief Title: Grip Effects of Power Ball in Children
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Riphah International University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Other
Other Study IDs: REC/RCR&AHS/23/0708
Record Dates: First submitted 2023-07-23; First posted 2023-08-04 (Actual); Last update posted 2023-11-13 (Actual); Status verified 2023-11

CONDITIONS: Visual Impairment
MeSH Terms: conditions — Vision Disorders

STUDY DESIGN:
Intervention Model Description: Its a randomized control trial,used to measure the grip strength of visually impared children by powerball.Subjects with visual impairment meeting the predetermined inclusion and exclusion criteria will be divided into two groups using random sampling technique
Who Masked: Participant
Masking Description: Participants will get separate tretment protocols and possible efforts will be put to mask the both groups about their treatment
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Conventional treatment of isometric hand grip training exercises (Active Comparator): In control group, conventional treatment perform by using isometric hand grip training exercises (putty grip and squeeze exercise, thumb pinch z strengthening exercises, isometric Hooks exercises, rubber band abduction and c thumb exercises) for 3times a week in one month.
  Interventions: Other: Conventional treatment of isometric hand grip training exercises
- Conventional treatment along with power ball training (Experimental): In experimental group, 3sessions per week and total 12 training sessions in a month will be perform. In this session, conventional treatment perform with power ball exercise should be done for 3 minutes in a day, where power ball can initially alleviate the pain, then make them feel strong and in the end persons feel strengthen with pain free movements. Before start training with a power ball, hand held dynamometer will use prior to the first session, on 7th session of training and after 12th training session. So that changes in hand grip strength can be measured by dynamometer.
  Interventions: Other: Conventional treatment along with power ball training

INTERVENTIONS:
Other: Conventional treatment of isometric hand grip training exercises — In control group, conventional treatment perform by using isometric hand grip training exercises (putty grip and squeeze exercise, thumb pinch z strengthening exercises, isometric Hooks exercises, rubber band abduction and c thumb exercises) for 3times a week in one month.
  Arms: Conventional treatment of isometric hand grip training exercises
Other: Conventional treatment along with power ball training — In experimental group, 3sessions per week and total 12 training sessions in a month will be perform. In this session, conventional treatment perform with power ball exercise should be done for 3 minutes in a day, where power ball can initially alleviate the pain, then make them feel strong and in the end persons feel strengthen with pain free movements. Before start training with a power ball, hand held dynamometer will use prior to the first session, on 7th session of training and after 12th training session. So that changes in hand grip strength can be measured by dynamometer.
  Arms: Conventional treatment along with power ball training

SUMMARY:
A broad definition of visual impairment includes a wide continuum of visual function loss. Aspects of visual function include visual acuity, which is the capacity to resolve detail, and accommodation (capacity to concentrate), field of vision (the area that may be seen), colour perception, and light sensitivity. A child with cerebral blindness can nevertheless be able to perceive motion. There are numerous sources of prevalence information, each of which has drawbacks. One of the fundamental pillars of the major worldwide prevention of blindness project, VISION 2020 the Right to Sight, is the reduction of visual impairment and blindness in children in resource-poor nations. Refraction and poor vision services aid visually impaired children, especially those with genetic or congenital ocular defects and enable vision improvement.

DETAILED DESCRIPTION:
Visual impairment is a broad term that describes a wide continuum of loss in visual function. There are many aspects of visual function e.g., visual acuity(ability to resolve detail),accommodation (ability to focus), field of vision (area which can be seen), colour vision and adapt ability to light. A child with cerebral blindness may have intact perception of movement. Prevalence data can be obtained from a variety of different sources, each of which has limitations. Reducing visual impairment and blindness in children in resource-poor countries is one of the key components of the major global prevention of blindness initiative, VISION 2020 the Right to Sight. Visually impaired children especially with hereditary /congenital ocular anomalies benefit from refraction and low vision services which facilitate vision enhancement and inclusive education. Pediatricians have a key role in early detection and multidisciplinary management to minimise the impact of visual impairment (VI) in childhood.Visually impaired children especially with hereditary /congenital ocular anomalies benefit from refraction and low vision services which facilitate vision enhancement and inclusive Powerball® is such a market existing device that can be used for wrist rehabilitation and also as a sports aid for strengthening the wrist. The Powerball acts as an eccentric exercise tool, generating forces in different directions and thus causing stimulation of the forearm, hand, and wrist musculature. The tools used will be handheld dynamometer and pegboard test. Study will be conducted on Twenty eight patients in two Groups. .Group A will be Control Group that will be provided with conventional physiotherapy (isometric hand grip training exercises) and Group B will be Experimental Group that Conventional treatment with power ball training. Data will be analyzed using spss 22.0

ELIGIBILITY:
Inclusion Criteria:

* Age ranging from 8 to 14 years,
* Both genders (male /female)

Exclusion Criteria:

* Serious medical conditions such as cardiac disease, diabetes, or uncontrolled seizures
* Significant shoulder, elbow, or
* wrist joint contractures preventing grip movement of the hand and fingers.
* Unable to follow the command
* Orthopedic surgery, neurological surgery

Ages: 8 Years to 14 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Enrollment: 30 (Actual)
Dates: Start 2023-07-15 (Actual); Primary Completion 2023-09-01 (Actual); Study Completion 2023-09-15 (Actual)

PRIMARY OUTCOMES:
Grip strength | 4 weeks
  grip strength will be meaured by dynamometer

SECONDARY OUTCOMES:
nine-hole peg test | 4 weeks
  nine-hole peg test will be utilized to measure grip performance..

CONTACTS AND LOCATIONS:
Overall Officials: Ahsan Taqweem, DPT, Principal Investigator — Riphah International University
Locations (1):
- Rising Sun Institute for Special Children, Lahore, Punjab Province, Pakistan

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Rasool J, Akram S, Jamil A, Tauseef M, Ilyas A. Effects of Power Ball Exercises in Addition to Routine Physical Therapy on Pain, Grip Strength and Functional Disability in Patients with Carpal Tunnel Syndrome: Power Ball Exercises in Carpal Tunnel Syndrome. The Healer Journal of Physiotherapy and Rehabilitation Sciences. 2023 May 3;3(4):451-60.